CLINICAL TRIAL: NCT06292065
Title: Gastric Ultrasound To Assess Gastric Contents In Patients On Semaglutide Therapy
Acronym: GUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nils Vlaeminck (Other)
Responsible Party: Sponsor-Investigator, Nils Vlaeminck, Principal investigator, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Project ID 6171
Record Dates: First submitted 2024-02-23; First posted 2024-03-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Intervention Model Description: 45 patients on semaglutide therapy will be included together with 45 age, BMI and diabetes status matched controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gastric Ultrasound (Experimental): Gastric ultrasound will be performed shortly before induction; i.e. in the preoperative room. The exam will be performed by the treating anaesthetist experienced with gastric ultrasound. The gastric antrum will be visualised in supine position followed by a second visualisation of the antrum in right lateral decubitus. In the latter position the cross-sectional area of the antrum (RIGHT-LAT CSA) will be measured and used to calculate the gastric volume using the [VOLUME (ML) = 27.0 + 14.6 X RIGHT-LAT CSA - 1.28 X AGE] formula. The patient will be considered to have a full stomach or positive gastric ultrasound if solid gastric content is visible in any visualisation of the antrum or if calculated liquid gastric content exceeds 1.5 ml/kg of total body weight.
  Interventions: Diagnostic Test: Point-of-care gastric ultrasound

INTERVENTIONS:
Diagnostic Test: Point-of-care gastric ultrasound — Using ultrasound to visualise the gastric antrum in supine position and right lateral decubitus.

SUMMARY:
Glucagon-like peptide-1 (GLP-1) receptor agonists (GLP-1-RA) such as semaglutide (Ozempic™, Rybelsus™, Wegovy™) were first introduced as a therapeutic agent for type 2 diabetes mellitus but they are being increasingly used to target weight loss in obesity.

One of the mechanisms by which weight loss is achieved, is increased satiety and significantly delayed gastric emptying. Tachyphylaxis for this effect has been reported with chronic use of long acting GLP-1-RA (e.g. semaglutide) but this was based on the paracetamol absorption technique or 13C breath test. Recent clinical data suggests semaglutide use does increase perioperative gastric content.This creates uncertainty for anaesthetists who are, anecdotally, more frequently faced with patients who may or may not have full stomachs despite adhering to conventional fasting guidelines.

To address this issue the American Society of Anesthesiologists (ASA) has recently released guidelines in which it advises to hold GLP-1-RA for one day (if administered daily) or one week (if administered weekly).

However, these recommendations are based on sparse empirical evidence and they do not necessarily follow from the known pharmacokinetic properties of these drugs. Typically, GLP-1-RA are administered in increasing doses over several weeks until a therapeutic steady state is achieved. Meanwhile the elimination half-life of e.g. semaglutide is 7 days. This means that holding semaglutide for one day or even one week might not be enough to attenuate its therapeutic effect of delayed gastric emptying. On the other hand if semaglutide were to be held for e.g. 5 terminal half-lifes, this would mean an unpractical 5 weeks during which glycemic control may be worsened and after which semaglutide doses would have to be incrementally increased again. Besides, hyperglycaemia secondary to semaglutide cessation can also delay gastric emptying.

Further confounding the assessment of these patients there can be 'background' delayed gastric emptying in diabetic patients and more pronounced delayed gastric emptying in patients recently started on GLP-1-RA. The presence of gastro-intestinal symptoms (nausea, vomiting, dyspepsia, abdominal distension) might offer clinical information regarding increased gastric residue in this population.

Gastric ultrasound is a point-of-care clinical and research tool that has steadily gained popularity to assess gastric content in patients not compliant with fasting rules or with certain comorbidities. Clinical decisions can be made based on the visualised content (e.g. solids, fluids or nothing) or through calculation of gastric volume by measuring antral circumference. In this study the investigators will examine gastric contents in patients who are taking semaglutide and in patients who are not. The investigators will then evaluate whether there is a difference in the incidence of full stomachs and whether gastric ultrasound influenced the anaesthetic plan of the treating anaesthetist.

ELIGIBILITY:
Inclusion criteria for the semaglutide cohort are:

* Adults (>=18 years old)
* Semaglutide therapy for any indication (type 2 diabetes or weight loss)
* Semaglutide therapy at any dose
* Semaglutide therapy with any route of administration
* Semaglutide therapy administered daily or weekly
* Semaglutide therapy at any time since initiation
* Elective surgery of any kind for which general anaesthesia was planned preoperatively
* Adherence to current ASA recommendation regarding GLP-1-RA; i.e. holding semaglutide for 1 week if administered weekly or for 1 day if administered daily.
* Adherence to current ESAIC fasting guidelines; i.e. >2 hours for liquids and >6 hours for solid foods.

Inclusion criteria for the control cohort are:

* Adults (>=18 years old)
* Elective surgery of any kind for which general anaesthesia was planned preoperatively
* Adherence to current ESAIC fasting guidelines; i.e. >2 hours for liquids and >6 hours for solid foods

Exclusion criteria for the semaglutide cohort are:

* Semaglutide not held in accordance with current ASA recommendation, i.e. held either longer or shorter than recommended.
* No adherence to current ESAIC fasting guideline
* Presence of a contra-indication to gastric ultrasound; i.e. previous gastric surgery (e.g. partial gastrectomy, gastric bypass) or hiatal hernias.
* Presence of comorbidities associated with delayed gastric emptying: scleroderma, systemic lupus erythematosus, hypothyroidism, Parkinson disease, cerebral palsy, and multiple sclerosis.
* Inability to assume the right lateral decubitus position
* Initial anaesthetic plan did not involve general anaesthesia, e.g. neuraxial or locoregional cases

Exclusion criteria for the control cohort are:

* Semaglutide or other GLP-1-RA therapy
* No adherence to current ESAIC fasting guideline
* Presence of a contra-indication to gastric ultrasound; i.e. previous gastric surgery (e.g. partial gastrectomy, gastric bypass) or hiatal hernias
* Presence of comorbidities associated with delayed gastric emptying: scleroderma, systemic lupus erythematosus, hypothyroidism, Parkinson disease, cerebral palsy, and multiple sclerosis
* Inability to assume the right lateral decubitus position
* Initial anaesthetic plan does not involve general anaesthesia, e.g. locoregional cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of full stomach | Immediately preoperatively
  The prevalence of a full stomach based on gastric ultrasound (solids visible in any visualisation or calculated liquid gastric content exceeding 1.5 ml/kg of total body weight) in patients taking semaglutide compared to controls

SECONDARY OUTCOMES:
Frequency of changes to the anaesthetic plan | Immediately preoperatively
  The frequency of changes to the anaesthetic plan (including postponement of surgery, change to locoregional or neuraxial technique, rapid sequence intubation, choice of airway, preoperative placement of nasogastric suctioning) after gastric ultrasound in semaglutide patients compared to controls
Calculated gastric content | Immediately preoperatively
  The calculated gastric content (median) based on gastric ultrasound in semaglutide patients compared to controls.
Prevalence of solid gastric content | Immediately preoperatively
  The prevalence of solid gastric content visible on gastric ultrasound in semaglutide patients compared to controls
Association between fasting time for solids and 'full stomach' | Immediately preoperatively
  The correlation between fasting time for solids and 'full stomach' on gastric ultrasound
Association between fasting time for liquids and 'full stomach' | Immediately preoperatively
  The correlation between fasting time for liquids and 'full stomach' on gastric ultrasound
Frequency of perioperative aspiration | Immediately postoperatively
  The frequency of perioperative aspiration of gastric contents in semaglutide patients compared to controls
Prevalence of gastric symptoms | Immediately preoperatively
  The prevalence of gastric symptoms (nausea, vomiting, dyspepsia, abdominal distension) in semaglutide patients compared to controls
Association between nausea and 'full stomach' | Immediately preoperatively
  The correlation between nausea and 'full stomach' on gastric ultrasound
Association between vomiting and 'full stomach' | Immediately preoperatively
  The correlation between vomiting and 'full stomach' on gastric ultrasound
Association between dyspepsia and 'full stomach' | Immediately preoperatively
  The correlation between dyspepsia and 'full stomach' on gastric ultrasound
Association between abdominal distension and 'full stomach' | Immediately preoperatively
  The correlation between abdominal distension and 'full stomach' on gastric ultrasound
association between semaglutide dose and calculated gastric content | Immediately preoperatively
  The correlation between semaglutide dose and calculated gastric content on gastric ultrasound
association between semaglutide dose and 'full stomach' | Immediately preoperatively
  The correlation between semaglutide dose and 'full stomach' on gastric ultrasound
Association between frequency of semaglutide administration and calculated gastric content | Immediately preoperatively
  The correlation between frequency of semaglutide administration and calculated gastric content on gastric ultrasound
Association between frequency of semaglutide administration and 'full stomach' | Immediately preoperatively
  The correlation between frequency of semaglutide administration and 'full stomach' on gastric ultrasound
Association between duration of semaglutide therapy and calculated gastric content | Immediately preoperatively
  The correlation between duration of semaglutide therapy and calculated gastric content on gastric ultrasound
Association between duration of semaglutide therapy at current dose and calculated gastric content | Immediately preoperatively
  The correlation between duration of semaglutide therapy at current dose and calculated gastric content on gastric ultrasound
Association between duration of semaglutide therapy and 'full stomach' | Immediately preoperatively
  The correlation between duration of semaglutide therapy and 'full stomach' on gastric ultrasound
Association between duration of semaglutide therapy at current dose and 'full stomach' | Immediately preoperatively
  The correlation between duration of semaglutide therapy at current dose and 'full stomach' on gastric ultrasound
Association between duration of cessation of semaglutide and calculated gastric content | Immediately preoperatively
  The correlation between duration of cessation of semaglutide therapy and calculated gastric content on gastric ultrasound in patients administering semaglutide daily and weekly
Association between duration of cessation of semaglutide and 'full stomach' | Immediately preoperatively
  The correlation between duration of cessation of semaglutide therapy and 'full stomach' on gastric ultrasound in patients administering semaglutide daily and weekly
Association between preoperative blood glucose levels and calculated gastric content | Immediately preoperatively
  The correlation between preoperative blood glucose levels and calculated gastric content on gastric ultrasound
Association between preoperative blood glucose levels and 'full stomach' | Immediately preoperatively
  The correlation between preoperative blood glucose levels and 'full stomach' on gastric ultrasound
Association between HbA1c levels and calculated gastric content | Immediately preoperatively
  The correlation between HbA1c levels and calculated gastric content on gastric ultrasound
Association between HbA1c levels and 'full stomach' | Immediately preoperatively
  The correlation between HbA1c levels and 'full stomach' on gastric ultrasound
Association between time since onset of diabetes mellitus and calculated gastric content | Immediately preoperatively
  The correlation between time since onset of diabetes mellitus and calculated gastric content on gastric ultrasound
Association between time since onset of diabetes mellitus and 'full stomach' | Immediately preoperatively
  The correlation between time since onset of diabetes mellitus and 'full stomach' on gastric ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Nils Vlaeminck, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No